CLINICAL TRIAL: NCT02770612
Title: Shared Decision Making for Prescription Opioids After Cesarean Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Brian Bateman, MD, MSc, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2016P000251
Record Dates: First submitted 2016-05-09; First posted 2016-05-12 (Estimated); Results first posted 2019-03-07 (Actual); Last update posted 2019-03-07 (Actual); Status verified 2019-03

CONDITIONS: Pregnancy; Cesarean Section; Prescriptions; Analgesics, Opioid

ARMS (1):
- Post-cesarean delivery mothers (Other): 1. Identify eligible women on post-operative day 3. A physician member of the study team will approach participants with study information and consent forms.
  2. After informed consent is obtained, the participant will be taken through a 10 minute shared decision making session (intervention). The participant will then have the opportunity to ask questions, following which they will indicate the number of prescription opioid tablets to be discharged with (primary outcome)
  3. The next contact will be at two weeks after discharge, at which time a member of the study team will contact the participant and administer a brief telephone survey with questions pertaining to perceived pain over time, pain management methods, opioid/pain medication consumption/disposal, and satisfaction with postoperative pain control.
  4. A chart review will be performed by physicians in the research group on participants to gather information on demographics, indications for surgery, etc.
  Interventions: Other: Prescribed opioids

INTERVENTIONS:
Other: Prescribed opioids — Making a shared decision with post-cesarean delivery mothers about quantity of opioids prescribed at discharge

SUMMARY:
The specific aim of this study is to use a shared decision making tool to allow women who have undergone cesarean delivery (CD) to choose the amount of oxycodone the participants will be prescribed at discharge, within a range from 0-40 tablets. The study investigators will document additional information from medical record abstraction (age, race/ethnicity, medical and obstetrical conditions, previous opioid use, date of CD, indication for CD, anesthetic management during CD, duration and complications of CD, length of stay, pain medication use and pain scores on each postoperative day between CD and discharge). The investigators will then follow up with the participants by telephone at two weeks after discharge to assess the amount of opioid used, frequency of prescription refill, disposition of unused medication, and participant satisfaction with their post-cesarean pain control. The investigators hypothesize that the use of a shared decision making tool will decrease the amount of opioid prescribed while still providing participants with satisfactory pain control.

ELIGIBILITY:
Inclusion Criteria:

* Postpartum women who underwent a cesarean delivery at MGH

Exclusion Criteria:

* Non-native English speakers (identified in LMR as "non-English speaking" or "requires interpreter")
* Women with a history of chronic opioid abuse (identified in LMR as "opioid abuse" or "narcotic abuse")
* Chronic pain on opioids (identified in LMR as "chronic pain" or "chronic narcotic use")
* Women on methadone or buprenorphine for treatment of opioid addiction (identified from their medication list in the LMR)
* Women with impaired decision-making abilities
* Women hospitalized for > 7 days related to CD
* Minors (<18 years old)
* Women being prescribed an opioid other than oxycodone during their postpartum hospitalization (identified from the MAR and discussion with rounding providers)
* Women with contraindications to taking acetaminophen or NSAIDs

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-04; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Prabhu M, McQuaid-Hanson E, Hopp S, Burns SM, Leffert LR, Landau R, Lauffenburger JC, Choudhry NK, Kaimal A, Bateman BT. A Shared Decision-Making Intervention to Guide Opioid Prescribing After Cesarean Delivery. Obstet Gynecol. 2017 Jul;130(1):42-46. doi: 10.1097/AOG.0000000000002094. PMID 28594762

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1 individual met exclusion criteria after agreeing to participate, due to postoperative length of stay > 7 days, and was not consented
Groups:
- Post-cesarean Delivery Mothers: Intervention: 10-minute shared decision making session via tablet
Period: Overall Study
Arm/Group | Post-cesarean Delivery Mothers
Started | 51
Completed | 50
Not Completed | 1
Not completed — Met exclusion criteria (postop LOS>7d) | 1

BASELINE CHARACTERISTICS:
Groups:
- Massachusetts General Hospital: Women who were postoperative day 3 from cesarean delivery, and were eligible Eligibility criteria
  1. English speaking
  2. using oral oxycodone
  3. age >=18
  4. post-operative length of stay less than 8 days
  5. no history of chronic pain or chronic opioid use
  6. lack of contraindications to tylenol/NSAIDs
Arm/Group | Massachusetts General Hospital
Number analyzed (Participants) | 50
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 33.0 [29.0 to 37.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 27
  Black | 0
  Hispanic | 8
  Asian | 14
  Other | 1
Type of cesarean delivery [Count of Participants; unit: Participants]
  Primary | 35
  Repeat | 15
Timing of cesarean delivery [Count of Participants; unit: Participants]
  Planned | 19
  Unplanned | 31
Postoperative length of stay [Median (Inter-Quartile Range); unit: days] | 4.0 [3.8 to 4.4]

OUTCOME MEASURES:

1. Primary Outcome: Pain Management and Opioid Usage Measured by Telephone Questionnaire
Description: Outpatient opioid selection and use after discharge
Time Frame: Within 2 weeks postpartum
Measure: Median (Inter-Quartile Range); unit: number of oxycodone 5mg tablets
Arm/Group | Massachusetts General Hospital
Number analyzed (Participants) | 50
number of oxycodone 5mg tablets
  Number of oxycodone tablets selected | 20.0 [15.0 to 25.0]
  Number of oxycodone tablets dispensed | 20.0 [20.0 to 30.0]
  Number of oxycodone tablets used | 15.5 [8.0 to 25.0]
  Number of oxycodone tablets remaining | 4.0 [0 to 8.0]
Statistical Analysis 1: Comparison: Massachusetts General Hospital; We used a one sided one sample Wilcoxon test to compare the median number of oxycodone tablets chosen and prescribed to the institutional standard of 40 tablets of oxycodone 5mg on discharge; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 2 weeks for each participant, as this was the timing of the post-discharge phone call
Groups:
- Post-cesarean Delivery Mothers: Women who were postoperative day 3 from cesarean delivery, and were eligible Eligibility criteria
  1. English speaking
  2. using oral oxycodone
  3. age >=18
  4. post-operative length of stay less than 8 days
  5. no history of chronic pain or chronic opioid use
  6. lack of contraindications to tylenol/NSAIDs
Arm/Group | Post-cesarean Delivery Mothers
All-Cause Mortality (participants affected / at risk) | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50
Other Adverse Events (participants affected / at risk) | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes